CLINICAL TRIAL: NCT07164313
Title: A First-In-Human, Phase 1, Open-Label, Multicenter Study of ZW251, a Novel Glypican-3 Targeting Antibody-Drug Conjugate, in Participants With Advanced Solid Tumors, Including Hepatocellular Carcinoma
Brief Title: A Study of ZW251 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zymeworks BC Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZWI-ZW251-101; 2025-523088-39 (EudraCT Number)
Record Dates: First submitted 2025-08-27; First posted 2025-09-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: GPC3-expressing cancer; hepatocellular carcinoma; antibody drug conjugate; ADC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZW251 (Experimental)
  Interventions: Drug: ZW251

INTERVENTIONS:
Drug: ZW251 — Administered intravenously

SUMMARY:
The purpose of this study is to find out if ZW251, an antibody-drug conjugate targeting glypican-3 (GPC3), is safe and can treat participants with advanced cancers, including hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Part 1 (dose escalation) of the study will evaluate the safety and tolerability of ZW251 in HCC. Part 2 (dose optimization) of the study will further assess safety and potential anti-tumor activity of the ZW251 established recommended doses in HCC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed diagnosis of HCC with evidence of locally advanced (unresectable, and ineligible for transplant) and/or metastatic disease. Noninvasive methods may be used to confirm diagnosis
* Measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Liver function status of Child-Pugh Class A
* Adequate organ function

Exclusion Criteria:

* Known additional malignancy that is progressing or that has required active treatment within the last year
* History of hepatic encephalopathy within the past 6 months or requirement for medications to control encephalopathy
* Portal vein thrombosis within 3 months prior to Cycle 1 Day 1 that require coagulation therapy or is not stable
* Known gastrointestinal bleeding within 3 months
* Acute or chronic uncontrolled renal disease, pancreatitis, or non-malignant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs; Part 1) | Up to 3 weeks
  Number of participants who experienced a DLT. DLTs include specifically defined adverse events (AEs) considered to be related to ZW251
Incidence of AEs (Parts 1 and 2) | Up to approximately 2 years
  Number of participants who experienced AEs, adverse events of special interest, or serious adverse events
Incidence of clinical laboratory abnormalities (Parts 1 and 2) | Up to approximately 2 years
  Number of participants who experienced a maximum severity of Grade 3 or higher post-baseline laboratory abnormality, including either hematology or chemistry. Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0
Confirmed objective response rate (Part 2) | Up to approximately 2 years
  Number of participants who achieved a best overall response of either confirmed complete response (CR) or partial response (PR) during treatment according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Confirmed objective response rate (Part 1) | Up to approximately 2 years
  Number of participants who achieved a best overall response of either confirmed CR or PR during treatment according to RECIST v1.1
Best overall response (Parts 1 and 2) | Up to approximately 2 years
Disease control rate (Parts 1 and 2) | Up to approximately 2 years
  Number of participants who achieved a best response of CR, PR, or stable disease during treatment per RECIST v1.1
Duration of response (Parts 1 and 2) | Up to approximately 2 years
  The time from the first objective response (CR or PR) to the first documented progressive disease (PD) per RECIST v1.1 or death within 30 days of last dose of study treatment from any cause. Only participants who achieve a confirmed response will be included in the analysis
Progression-free survival (Parts 1 and 2) | Up to approximately 2 years
  The time from the first dose of study treatment to the date of first documented PD per RECIST v1.1 or death from any cause
Overall survival (Part 2) | Up to approximately 2 years
  The time from the date of the first dose of study treatment to the date of death due to any cause
Area under the concentration-time curve (AUC0-504) of ZW251 (Parts 1 and 2) | Up to approximately 2 years
  Area under the concentration-time curve of ZW251 after first dose administration
Maximum concentration (Cmax) of ZW251 (Parts 1 and 2) | Up to approximately 2 years
  ZW251 maximum concentration after first dose administration
Area under the concentration-time curve of ZW251 at steady state (AUCtau,ss; Parts 1 and 2) | Up to approximately 2 years
  Area under the concentration-time curve of ZW251 at steady state after fourth dose administration
Maximum concentration of ZW251 at steady state (Сmax,ss; Parts 1 and 2) | Up to approximately 2 years
  ZW251 maximum concentration at steady state after fourth dose administration
Minimal concentration of ZW251 at steady state (Сmin,ss; Parts 1 and 2) | Up to approximately 2 years
  ZW251 minimal concentration at steady state after fourth dose administration
Incidence of anti-drug antibodies (ADAs; Parts 1 and 2) | Up to approximately 2 years
  Number of participants who develop ADAs

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Weinstein, MD, PhD, MPH, Study Director — Zymeworks BC Inc.
Locations (10):
- United States (5):
  - Norton Cancer Institute, Louisville, Kentucky
  - START Midwest, Grand Rapids, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - MD Anderson Cancer Center, Houston, Texas
  - START San Antonio, San Antonio, Texas
- Japan (3):
  - Kyoto University Hospital, Kyoto
  - Kansai Medical University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No